CLINICAL TRIAL: NCT01712204
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Of AC-201 In Subjects With Gout Initiating Urate-Lowering Therapy
Brief Title: A Proof-of-Concept Study of AC-201 to Prevent Gout Flares
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TWi Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AC-201-GOU-001
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Gout Flares
Keywords: Prophylaxis of Acute Gout Flares; Urate-Lowering Therapy; Hyperuricemia; Gouty arthritis
MeSH Terms: conditions — Hyperuricemia; Arthritis, Gouty | interventions — diacerein; Febuxostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo plus Febuxostat
  Interventions: Drug: Placebo; Drug: Febuxostat
- AC-201 (Experimental): AC-201 plus Febuxostat
  Interventions: Drug: AC-201; Drug: Febuxostat

INTERVENTIONS:
Drug: Placebo — Placebo Capsule BID for 16 Weeks
  Other Names: PBO
  Arms: Placebo
Drug: AC-201 — AC-201 50mg Capsule BID for 16 Weeks
  Arms: AC-201
Drug: Febuxostat — Febuxostat 80 mg QD for 16 Weeks
  Other Names: ULT

SUMMARY:
Initiation of ULT for gout increases the occurrence of acute gouty arthritis flares due to mobilization of urate from tissue deposits. IL-1β plays a key role in mediating the inflammatory response in gouty arthritis. The efficacy of IL-1β blockade in the prophylaxis of gouty flares during initiation of ULT has been validated in multiple trials of IL-1β inhibitor therapies. Therefore, it is believed that IL-1β is a relevant therapeutic target for gout flares. AC-201 is an IL-1β modulator indicated for the treatment of osteoarthritis with good safety record and very few contraindications to the co-morbidities commonly among gout patients. AC-201 has also been demonstrated to have uric acid-lowering effects in clinical trials. The favorable product profile of AC-201 overall provides a strong rationale for investigating its clinical utility as prophylaxis against flares when initiating ULT.

DETAILED DESCRIPTION:
Clinical trials have demonstrated that anti-IL-1 agents (IL-1Ra, IL-1 Trap, and anti-IL-1β monoclonal antibody) can reduce the frequency of gout flares during the initial period of treatment with urate-lowering therapy and prevent of gout flares in gout patients with frequent flares. AC-201 is an oral IL-1 modulator but with a mechanism distinct from that of existing anti-IL-1 agents. The active metabolite of AC-201 has been shown in vitro and in vivo to inhibit the production and activity of IL-1, down-regulate IL-1 receptors, and increase IL1-Ra. Molecular research further suggests that these effects are mediated upstream via inhibition of MAPK signaling pathways and binding of NF-κB and AP-1 transcription factors that encode for a range of pro-inflammatory factors, including IL-1β, TNF-α, IL-6, IL-8, iNOS, and MMPs, which have been implicated in gout flares. AC-201 has also been demonstrated to have uric acid-lowering effects in clinical trials. The favorable product profile of AC-201 overall provides a strong rationale for investigating its clinical utility as prophylaxis against flares when initiating ULT.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 20 to 80 years, inclusive
* Meets at least 6 of the 12 American College of Rheumatology preliminary criteria (1977) for the classification of acute arthritis of primary gout, OR have proven tophus or documented monosodium urate (MSU) crystals in the joint fluid
* Serum uric acid ≥7.5 mg/dL at screening
* Experienced ≥2 gouty arthritis flares within one year prior to screening

Exclusion Criteria:

* Occurrence of a gouty arthritis flare ongoing at screening or during the screening period through baseline
* Use of allopurinol, febuxostat, benzbromarone, probenecid, or sulfinpyrazone within 4 weeks prior to screening
* Use of colchicine, glucocorticoids, NSAIDs, or COX-2 inhibitors within 1 week prior to screening
* Other (non-gout) chronic arthritis, acute inflammatory arthritis, autoimmune diseases with arthritis, or any condition requiring chronic daily use of pain medication
* History of allergy to any components of study medication, including diacerein
* Allergy, contraindication, or intolerance to febuxostat
* Contraindication or allergy to NSAIDs
* Severe renal impairment
* Any prior use of biologic anti-inflammatory therapy, such as IL-1 modulators, tumor necrosis factor inhibitors, IL-6 inhibitors, or T-cell costimulation modulator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Veterans General Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 82 patients from 8 clinical centers participated in the study between 28 January 2013 to 04 September 2013.
Pre-assignment Details: Participants were assessed at an initial screening visit within 2 weeks before the baseline visit.
Period: Overall Study
Arm/Group | Placebo | AC-201
Started | 41 | 41
Completed | 33 | 36
Not Completed | 8 | 5
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: A total of 82 subjects were randomized and received at least one dose of study medication (the Intent-to-Treat [ITT] Population). The ITT Population was used for baseline/demographic, disposition, and safety summaries. The ITT Population was the primary analysis set for efficacy analyses.
Groups:
- Placebo Capsule BID: Placebo Capsule BID for 16 Weeks
- AC-201 50mg Capsule BID: AC-201 50mg Capsule BID for 16 Weeks
- Total: Total of all reporting groups
Arm/Group | Placebo Capsule BID | AC-201 50mg Capsule BID | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (11.8) | 43.7 (12.6) | 43.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 41 | 41 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Gout Flares Per Subject
Time Frame: 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: flares
Groups:
- Placebo: Placebo Capsule BID for 16 Weeks
  Background therapy: Urate-Lowering Therapy (Febuxostat 80 mg QD)
- AC-201: AC-201 50mg Capsule BID for 16 Weeks
  Background therapy: Urate-Lowering Therapy (Febuxostat 80 mg QD)
Arm/Group | Placebo | AC-201
Number analyzed (Participants) | 41 | 41
flares | 3.02 [2.51 to 3.64] | 2.45 [2.01 to 3.00]
Statistical Analysis 1: Comparison: Placebo vs AC-201; Test type: Superiority or Other; p = 0.1356, Possion regression; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.62 to 1.07], Standard Error of Mean 0.113

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Placebo | AC-201
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/41
Other Adverse Events (participants affected / at risk) | 11/41 | 10/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=41) | AC-201 (N=41)
Frequent Gout Attack (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=41) | AC-201 (N=41)
Blood CPK increased (Investigations) | 4 (4) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 2 (2)
ALT increased (Investigations) | 3 (3) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less